CLINICAL TRIAL: NCT05967637
Title: The Effect of Whole-Body Vibration Treatment Before Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sevim Beyza Ölmez, Principal Investigator, PhD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-874
Record Dates: First submitted 2023-07-11; First posted 2023-08-01 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Whole-body Vibration; Arthropathy of Knee; Swelling/ Edema
Keywords: whole-body vibration; total knee arthroplasty; swelling; edema
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-body vibration (Experimental): Standard patient education and exercise training + whole body vibration
  Interventions: Other: Whole body vibration
- Sham-whole-body vibration (Sham Comparator): Standard patient education and exercise training + sham whole body vibration
  Interventions: Other: Sham-Whole body vibration

INTERVENTIONS:
Other: Whole body vibration — The vibration will be applied for 10 minutes (30 seconds rest, 30 seconds training, 10 reps) in total with a low frequency (20 HZ) and low amplitude (2mm). Participants will be asked to stand in a squatting position by semi-flexing (30°) their knees during the 30-second vibration period.
  Arms: Whole-body vibration
Other: Sham-Whole body vibration — The sham-whole body vibration treatment will follow the same procedures with the vibration machine off.
  Arms: Sham-whole-body vibration

SUMMARY:
The study's objective is to investigate the effects of whole-body vibration therapy administered before surgery on various factors related to patients who undergo total knee arthroplasty. These factors include pain, swelling, skin temperature, normal joint movement, knee joint position sense, knee extensor muscle strength, functional status, and patient satisfaction.

DETAILED DESCRIPTION:
The study will include participants aged 50-80 who are planning to undergo total knee arthroplasty. According to the sample size analysis, a total of 40 people will be included in this study. The enrolled participants will be randomly assigned to one of two parallel groups: the whole-body vibration group or the sham whole-body vibration group. Both groups will receive standard patient education and exercise training.The experimental group will receive whole-body vibration along with exercise on the whole-body vibration device, while the control group (sham group) will receive sham vibration on the same device. All participants will receive treatment for a total of 5 days, one session per day.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced idiopathic knee OA and scheduled for unilateral total knee arthroplasty will be considered candidates for the present study and will be asked to participate

Exclusion Criteria:

* if they had undergone another hip or knee joint replacement in the previous year
* if they had any medical condition in which exercise was contraindicated
* if they had any disease that affected functional performance

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Baseline pain severity | baseline
  The pain severity will be evaluated using an NRS rating from 0 to 10, with 0 representing no pain and 10 representing maximal pain.
Change in pain severity from baseline to day 5 after interventions | up to 5 days after baseline
  The pain severity will be evaluated using an NRS rating from 0 to 10, with 0 representing no pain and 10 representing maximal pain.pain and 10 representing maximal pain.
Change in the preoperative pain severity on the 7th day of surgery | up to 7 days after surgery
  The pain severity will be evaluated using an NRS rating from 0 to 10, with 0 representing no pain and 10 representing maximal pain.
Change in pain severity from day 7 to day 14 post-surgery | up to 14 days after surgery
  The pain severity will be evaluated using an NRS rating from 0 to 10, with 0 representing no pain and 10 representing maximal pain.
Change in pain severity from day 14 to day 21 post-surgery | up to 21 days after surgery
  The pain severity will be evaluated using an NRS rating from 0 to 10, with 0 representing no pain and 10 representing maximal pain.
Baseline leg circumference | baseline
  Knee swelling will be assessed by measuring the circumference of the mid-patella, thigh, and calf with the knee in full extension.
Change in leg circumference from baseline to day 5 after interventions | up to 5 days after baseline
  Knee swelling will be assessed by measuring the circumference of the mid-patella, thigh, and calf with the knee in full extension.
Change in the preoperative leg circumference on the 7th day of surgery | up to 7 days after surgery
  Knee swelling will be assessed by measuring the circumference of the mid-patella, thigh, and calf with the knee in full extension.
Change in leg circumference from day 7 to day 14 post-surgery | up to 14 days after surgery
  Knee swelling will be assessed by measuring the circumference of the mid-patella, thigh, and calf with the knee in full extension.
Change in leg circumference from day 14 to day 21 post-surgery | up to 21 days after surgery
  Knee swelling will be assessed by measuring the circumference of the mid-patella, thigh, and calf with the knee in full extension.
Baseline range of motion | baseline
  The knee flexion and extension ranges of motion will be measured using a goniometer in the supine position.
Change in range of motion from baseline to day 5 after interventions | up to 5 days after baseline
  The knee flexion and extension ranges of motion will be measured using a goniometer in the supine position.
Change in the preoperative range of motion on the 7th day of surgery | up to 7 days after surgery
  The knee flexion and extension ranges of motion will be measured using a goniometer in the supine position.
Change in range of motion from day 7 to day 14 post-surgery | up to 14 days after surgery
  The knee flexion and extension ranges of motion will be measured using a goniometer in the supine position.
Change in range of motion from day 14 to day 21 post-surgery | up to 21 days after surgery
  The knee flexion and extension ranges of motion will be measured using a goniometer in the supine position.
Baseline muscle strength | baseline
  Knee extensor muscle strength will be assessed using a hand-held dynamometer in the sitting position.
Change in muscle strength from baseline to day 5 after interventions | up to 5 days after baseline
  Knee extensor muscle strength will be assessed using a hand-held dynamometer in the sitting position.
Change in the preoperative muscle strength on the 7th day of surgery | up to 7 days after surgery
  Knee extensor muscle strength will be assessed using a hand-held dynamometer in the sitting position.
Change in muscle strength from day 7 to day 14 post-surgery | up to 14 days after surgery
  Knee extensor muscle strength will be assessed using a hand-held dynamometer in the sitting position.
Change in muscle strength from day 14 to day 21 post-surgery | up to 21 days after surgery
  Knee extensor muscle strength will be assessed using a hand-held dynamometer in the sitting position.
Baseline skin temperature | baseline
  A portable infrared thermometer will be used to measure knee skin temperature.
Change in skin temperature from baseline to day 5 after interventions | up to 5 days after baseline
  A portable infrared thermometer will be used to measure knee skin temperature.
Change in the preoperative skin temperature on the 7th day of surgery | up to 7 days after surgery
  A portable infrared thermometer will be used to measure knee skin temperature.
Change in skin temperature from day 7 to day 14 post-surgery | up to 14 days after surgery
  A portable infrared thermometer will be used to measure knee skin temperature.
Change in skin temperature from day 14 to day 21 post-surgery | up to 21 days after surgery
  A portable infrared thermometer will be used to measure knee skin temperature.
Baseline knee proprioception | baseline
  Active reposition test will be measured using a digital inclinometer device.
Change in knee proprioception from baseline to day 5 after interventions | up to 5 days after baseline
  Active reposition test will be measured using a digital inclinometer device.
Change in the preoperative knee proprioception on the 7th day of surgery | up to 7 days after surgery
  Active reposition test will be measured using a digital inclinometer device.
Change in knee proprioception from day 7 to day 14 post-surgery | up to 14 days after surgery
  Active reposition test will be measured using a digital inclinometer device.
Change in knee proprioception from day 14 to day 21 post-surgery | up to 21 days after surgery
  Active reposition test will be measured using a digital inclinometer device.
Baseline Time Up and Go | baseline
  functional performance test
Change in Time Up and Go from baseline to day 5 after interventions | up to 5 days after baseline
  functional performance test
Change in the preoperative Time Up and Go on the 7th day of surgery | up to 7 days after surgery
  functional performance test
Change in Time Up and Go from day 7 to day 14 post-surgery | up to 14 days after surgery
  functional performance test
Change in Time Up and Go from day 14 to day 21 post-surgery | up to 21 days after surgery
  functional performance test

SECONDARY OUTCOMES:
SF-36 | baseline
  The 36-Item Short-Form Health Survey (SF-36) is a general scoring instrument used to provide a health profile comprised of eight scaled scores. Each scale is instantly turned into a 0-100 scale, allowing identification of the patient's physical and mental status. A higher score means a better result.
Change in the preoperative SF-36 on the 21st day of surgery | up to 21 days after surgery
  The 36-Item Short-Form Health Survey (SF-36) is a general scoring instrument used to provide a health profile comprised of eight scaled scores. Each scale is instantly turned into a 0-100 scale, allowing identification of the patient's physical and mental status. A higher score means a better result.
WOMAC | before interventions, 21st day after surgery
  The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a disease-specific self-report multidimensional questionnaire that assesses pain, stiffness, and physical functional disability. A higher score means a better result.
Change in the preoperative WOMAC on the 21st day of surgery | up to 21 days after surgery
  The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a disease-specific self-report multidimensional questionnaire that assesses pain, stiffness, and physical functional disability. A higher score means a better result.
Global Rating of Change Scales (GROC) | up to 21st day after surgery
  The GROC score, which has seven response options ranging from 'much worse' (a score of 0) to 'much better' (a score of six), will be used to determine the subject's perception of overall improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Hazar, Study Director — Gazi University; Cemil Yıldız, Study Chair — Gulhane Training and Research Hospital; Sevim Beyza Ölmez, Principal Investigator — Gazi University; Beyza Yazgan, Principal Investigator — Gazi University; İnci Ayaş, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No